CLINICAL TRIAL: NCT06394778
Title: Electroencephalogram Characteristics of Surgical Anesthetized Patients and Their Correlation With Postoperative Delirium
Brief Title: Electroencephalogram Characteristics of Surgical Anesthetized Patients and Postoperative Dilirium
Status: Enrolling by invitation | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Gan Shuyuan, associate chief physician, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20240135B-R1
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Electroencephalogram; Postoperative Delirium (POD)
Keywords: Single-center, prospective, observational, case-control study
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium group: If the patient develops delirium after surgery, he/she is in the delirium group
  Interventions: Diagnostic Test: Delirium test scale：3D-CAM
- Non delirium group: If the patient does not experience delirium after surgery, it is considered as the non-delirium group
  Interventions: Diagnostic Test: Delirium test scale：3D-CAM

INTERVENTIONS:
Diagnostic Test: Delirium test scale：3D-CAM — The 3D-CAM is a 3-minute delirium assessment that is also based upon the CAM algorithm and has four features: (1) altered mental status/fluctuating course, (2) inattention, (3) altered level of consciousness, and (4) disorganized thinking.

SUMMARY:
Objective: To construct a perioperative EEG database for elderly patients under general anesthesia and to explore the relationship between their EEG spectrum characteristics and the occurrence and severity of postoperative delirium. Content: This study aims to investigate elderly patients undergoing elective orthopedic surgery under general anesthesia with endotracheal intubation, analyze the changes in the perioperative EEG spectrum and its correlation with the occurrence of postoperative delirium, and explore the relationship between perioperative EEG changes and the occurrence of postoperative delirium. Methods: Patients aged 60 years or older who were scheduled to undergo orthopedic joint replacement or spinal surgery and had a hospital stay of more than 2 days were selected. All patients underwent MMSE and 3D-CAM assessment before surgery. Before anesthesia induction, anesthesia depth monitoring electrodes were placed on the patient's occipital or frontal temporal region, and EEGs were collected in awake and quiet states, under general anesthesia, and during anesthesia recovery. In the PACU, the score was calculated based on the CAM-ICU scale. The patients were assessed with the 3D-CAM scale for awakening once a day at 15:00-20:00 the day before surgery, and twice a day at 9:00-11:00 and 15:00-20:00 during 1-5 days after surgery, or at any time when obvious delirium symptoms appeared, unless discharged from the hospital or taking sedatives (RASS<-3). Ten minutes after the assessment, the occipital EEG was monitored when the patient was conscious and quiet, or when obvious delirium appeared. According to the test results of the 3D-CAM scale, it was determined whether the patient had postoperative delirium, and the patients were divided into the delirium group and the non-delirium group. The EEG characteristics of the two groups of patients were analyzed before, during, and after surgery. Research significance: The results of this study can provide objective indicators and theoretical basis for monitoring and diagnosing the occurrence and development of POD, which can help clinicians to identify patients with increased risk of delirium at an early stage, adjust the plan in time, and change the triggering risk factors of POD.

DETAILED DESCRIPTION:
Preoperative cognitive and delirium assessment:

MMSE scale assesses the patient's preoperative cognitive function status: the total score is 30 points, the higher the score, the better the cognitive function. Considering the impact of education level on MMSE assessment, combined with my country's actual situation and previous studies, we set the assessment criteria for illiterate or most primary and junior high school education levels to ≤17, ≤20, and ≤24, respectively. Individuals below the corresponding standards are considered to have cognitive impairment before surgery.

Preoperative 3D-CAM baseline value for delirium assessment: patients were assessed for delirium using the 3-minute rapid mental confusion assessment method (3D-CAM) between 15:00 and 20:00 the day before surgery.

Postoperative delirium assessment:

During the postoperative PACU period, the score was calculated based on the CAM-ICU scale; 1-5 days after surgery, patients underwent 3D-CAM assessment twice a day at 9:00-11:00 and 15:00-20:00, or at any time when obvious delirium symptoms appeared, unless discharged or taking sedatives (RASS<-3).

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 60 years, scheduled for orthopedic joint replacement or spinal surgery, ASA grade I-III, expected surgery time ≥ 2 hours, and able to provide written informed consent.

Exclusion Criteria:

1. Patients with central nervous system diseases or mental disorders;
2. patients with severe systemic diseases such as cardiopulmonary, liver and kidney dysfunction, coagulation dysfunction, etc.;
3. patients who frequently use psychotropic drugs, opioids or corticosteroids;
4. patients with a history of intraoperative awareness;
5. patients who are unable to complete preoperative delirium screening due to severe blindness, deafness, illiteracy or Mandarin speaking;
6. patients who are expected to undergo a second operation within 7 days.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients undergoing elective orthopedic joint replacement or spinal surgery
Sampling Method: Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between perioperative EEG spectral changes and postoperative delirium | 2 years
  Characteristic changes of EEG spectral changes in patients with POD before, during, and after surgery
Incidence of POD | 1 years
  The proportion of POD occurrence

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ravi B, Pincus D, Choi S, Jenkinson R, Wasserstein DN, Redelmeier DA. Association of Duration of Surgery With Postoperative Delirium Among Patients Receiving Hip Fracture Repair. JAMA Netw Open. 2019 Feb 1;2(2):e190111. doi: 10.1001/jamanetworkopen.2019.0111. PMID 30794305
- [Result] Gan S, Yu Y, Wu J, Tang X, Zheng Y, Wang M, Zhu S. Preoperative assessment of cognitive function and risk assessment of cognitive impairment in elderly patients with orthopedics: a cross-sectional study. BMC Anesthesiol. 2020 Aug 1;20(1):189. doi: 10.1186/s12871-020-01096-6. PMID 32738902
- [Result] Kinoshita H, Saito J, Kushikata T, Oyama T, Takekawa D, Hashiba E, Sawa T, Hirota K. The Perioperative Frontal Relative Ratio of the Alpha Power of Electroencephalography for Predicting Postoperative Delirium After Highly Invasive Surgery: A Prospective Observational Study. Anesth Analg. 2023 Dec 1;137(6):1279-1288. doi: 10.1213/ANE.0000000000006424. Epub 2023 Mar 14. PMID 36917508
- [Result] Koch S, Windmann V, Chakravarty S, Kruppa J, Yurek F, Brown EN, Winterer G, Spies C; BioCog Study Group. Perioperative Electroencephalogram Spectral Dynamics Related to Postoperative Delirium in Older Patients. Anesth Analg. 2021 Dec 1;133(6):1598-1607. doi: 10.1213/ANE.0000000000005668. PMID 34591807
- [Result] Hesse S, Kreuzer M, Hight D, Gaskell A, Devari P, Singh D, Taylor NB, Whalin MK, Lee S, Sleigh JW, Garcia PS. Association of electroencephalogram trajectories during emergence from anaesthesia with delirium in the postanaesthesia care unit: an early sign of postoperative complications. Br J Anaesth. 2019 May;122(5):622-634. doi: 10.1016/j.bja.2018.09.016. Epub 2018 Oct 25. PMID 30915984
- [Result] Lutz R, Muller C, Dragovic S, Schneider F, Ribbe K, Anders M, Schmid S, Garcia PS, Schneider G, Kreuzer M, Kratzer S. The absence of dominant alpha-oscillatory EEG activity during emergence from delta-dominant anesthesia predicts neurocognitive impairment- results from a prospective observational trial. J Clin Anesth. 2022 Nov;82:110949. doi: 10.1016/j.jclinane.2022.110949. Epub 2022 Aug 29. PMID 36049381
- [Result] Boord MS, Moezzi B, Davis D, Ross TJ, Coussens S, Psaltis PJ, Bourke A, Keage HAD. Investigating how electroencephalogram measures associate with delirium: A systematic review. Clin Neurophysiol. 2021 Jan;132(1):246-257. doi: 10.1016/j.clinph.2020.09.009. Epub 2020 Oct 1. PMID 33069620
- [Result] Kassie GM, Nguyen TA, Kalisch Ellett LM, Pratt NL, Roughead EE. Preoperative medication use and postoperative delirium: a systematic review. BMC Geriatr. 2017 Dec 29;17(1):298. doi: 10.1186/s12877-017-0695-x. PMID 29284416
- [Result] Kaiser HA, Peus M, Luedi MM, Lersch F, Krejci V, Reineke D, Sleigh J, Hight D. Frontal electroencephalogram reveals emergence-like brain activity occurring during transition periods in cardiac surgery. Br J Anaesth. 2020 Sep;125(3):291-297. doi: 10.1016/j.bja.2020.05.064. Epub 2020 Jul 15. PMID 32682555
- [Result] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Result] Tsai MC, Chou SY, Tsai CS, Hung TH, Su JA. Comparison of consecutive periods of 1-, 2-, and 3-year mortality of geriatric inpatients with delirium, dementia, and depression in a consultation-liaison service. Int J Psychiatry Med. 2013;45(1):45-57. doi: 10.2190/PM.45.1.d. PMID 23805603
- [Result] Jabbar F, Leonard M, Meehan K, O'Connor M, Cronin C, Reynolds P, Meaney AM, Meagher D. Neuropsychiatric and cognitive profile of patients with DSM-IV delirium referred to an old age psychiatry consultation-liaison service. Int Psychogeriatr. 2011 Sep;23(7):1167-74. doi: 10.1017/S1041610210002383. Epub 2011 Jan 21. PMID 21251353
- [Result] Blazer DG, van Nieuwenhuizen AO. Evidence for the diagnostic criteria of delirium: an update. Curr Opin Psychiatry. 2012 May;25(3):239-43. doi: 10.1097/YCO.0b013e3283523ce8. PMID 22449764